CLINICAL TRIAL: NCT00194974
Title: Treatment Targets for Chronic Hypertension in Pregnancy
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0304-191
Record Dates: First submitted 2005-09-13; First posted 2005-09-19 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2017-01

CONDITIONS: Pregnancy Toxemia; Hypertension; Proteinuria
Keywords: pregnancy; chronic hypertension; Toxemia; Blood Pressure
MeSH Terms: conditions — Pre-Eclampsia; Hypertension; Proteinuria; Toxemia | interventions — Methyldopa; Labetalol; Nifedipine; Clonidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: methyldopa
Drug: labetalol
Drug: nifedipine
Drug: clonidine

SUMMARY:
This project is a clinical study of women with high blood pressure who become pregnant. Preeclampsia is a syndrome developing at the end of a pregnancy characterized by an abrupt rise in blood pressure (BP), blood clotting and kidney dysfunction, and may result in premature delivery, infant death, and maternal bleeding, kidney failure and stroke. The goal is to determine whether lowering blood pressure to a normal pressure of 120/80 is associated with a lower incidence of preeclampsia. Women who are completely healthy have a 5% chance of developing preeclampsia, however women with preexisting high blood pressure have a 25% chance of this complication. Several studies, including our own suggest that higher blood pressure early in pregnancy (<20 weeks) is associated with an even higher risk of preeclampsia. Currently we, the researchers at Weill Medical College of Cornell University, do not know how to treat women with high blood pressure and/or kidney disease during pregnancy. Keeping the BP in the normal range may be beneficial to the mother. On the other hand, we are not sure if the blood pressure lowering or the medications may or may not have adverse effects for the baby. Different trials to answer this question have been performed with no clear conclusions. Because of these uncertainties, we propose to compare two different strategies for treating women with high BP who become pregnant. We will treat half the women with BP medications to normalize BP (120-130/80 mm Hg) (experimental group) and the other half with the goal of keeping the BP slightly higher (140-150/90-100 mm Hg)(standard therapy group). We will determine which approach results in healthier pregnancies, and lower incidence of preeclampsia. Reducing the incidence of preeclampsia would be of significant benefit to both mothers and babies.

DETAILED DESCRIPTION:
Methods:

This is a pilot study to examine the feasibility of conducting a larger, multi center randomized control trial. Fifty women with chronic hypertension who are pregnant and are seen in the first trimester of pregnancy will be recruited from the offices of obstetricians at New York Presbyterian Hospital.

Recruitment:

First trimester (up to 13 6/7th weeks)

Stratified by:

* Parity (primiparous vs. multiparous delivering a fetus >20 weeks gestation)
* Severity of hypertension (>150/95) as determined on screening antepartum visit

Inclusion Criteria:

1. Pregnant patients will be evaluated for recruitment to 13 6/7 weeks gestation.
2. Age 18-50
3. Patients will be included for consideration to enter this trial if office blood pressure is >140/90 mm Hg: systolic >140 mm Hg, diastolic >90 mm Hg or both. The average of 3 readings taken a minimum of 5 minutes apart will be recorded as the baseline blood pressure.
4. Patients will also be included for consideration to enter this trial if they have known longstanding hypertension diastolic blood pressure (DBP) >90 within 2 years of index pregnancy and/or are on antihypertensive medication, regardless of in-office blood pressure if seen in their first trimester.

Exclusion Criteria:

Significant target organ damage; at the patient's initial antepartum visit, routine serum creatinine and urine dipstick for protein are performed by the attending obstetrician. If the patient has been hypertensive by history for over 5 years, a screening electrocardiogram will be performed. These will be reviewed for results precluding participation in the trial.

1. Known renal disease creatinine > 1.2 mg/dl
2. Proteinuria >500 mg/day at baseline
3. Left ventricular hypertrophy by electrocardiography (ECG) criteria.
4. History of the following: chronic illness requiring immunosuppression, as well as secondary causes of hypertension: pheochromocytoma, hyperaldosteronism, coarctation of aorta, renal artery stenosis not revascularized.

NB: the presence of the above conditions would make it more likely that a clinician would treat blood pressure during pregnancy. Therefore, the patient may be randomized and treatment begun as per protocol prior to complete evaluation of presence of above conditions; if exclusion criteria are subsequently identified the patient would then be excluded and treated according to individual physicians standard of practice.

Enrollment:

Patients will undergo initial baseline evaluation. History and physical will be performed. Weight, height and blood pressure will be recorded.

Eligible patients will sign informed consent. Each patient will have a data sheet for the purpose of recording study results.

Randomization:

Patients will be randomized to one of two blood pressure targets:

120-130/80-85 mm Hg vs. 140-150/90-100 mm Hg

Randomization will occur by blocked randomization in blocks of 6. Randomization is stratified for parity (nulliparous vs. multiparous) and severe vs. non-severe hypertension. There are therefore 4 potential groups:

1. Nulliparous + non-severe hypertension
2. Multiparous + non-severe hypertension
3. Nulliparous + severe hypertension
4. Multiparous + severe hypertension

There are 54 envelopes for each group (allowing for the theoretic possibility that all patients may fall into one group) and envelopes are numbered and will be opened sequentially to allocate patients during the randomization process.

Treatment:

Patients with no prior history of hypertension will be treated as per the protocol described below.

Patients with a known history of hypertension will still be randomized to the appropriate group according to parity and blood pressure in clinic, but will be asked to stop their antihypertensive medication for a wash out period.

The patient will then return to clinic three to seven days later off medication to have a repeat blood pressure measurement. If they own a home blood pressure monitor and this has been calibrated to office equipment, they may take their blood pressure at home.

They will be then be treated as per their randomization group i.e. to a blood pressure of 120-130/80-85 mm Hg vs. 140-150/90-100 mm Hg as per the protocol below.

The patient will be given a diary to record obstetric data and blood pressure data. Duplicate records will be kept by the patient and physician.

Weight, blood pressure, pulse, presence or absence of edema and urinary protein will be recorded at each visit.

Medication Protocol:

Treatment is to commence immediately after randomization unless the patient is undergoing a washout period described above.

Some patients will initially require no medication as BP's may be below the treatment threshold, depending on their treatment group.

Treatment will be with methyldopa, labetolol, long acting nifedipine, hydralazine or clonidine.

Scheduled Visits:

Patients will be followed every two to four weeks until delivery. Medication will be titrated to achieve the desired blood pressure targets. Patients will not be billed for these visits.

The achievement of target blood pressure will be assessed by an average of three blood pressure measurements obtained at every six weeks visits: weeks 20, 26, 32 and 38.

At the 20 week visit, routine blood work will be drawn to evaluate uric acid and plasma renin activity as validation of the prediction algorithm.

Home Blood Pressure Monitoring:

If patients own a home blood pressure monitor, they will be asked to bring it into clinic for calibration. They will be given a blood pressure diary to record home blood pressure monitoring or BP measurements done in another clinic or pharmacy.

Duration of Treatment:

The treatment goals of 120-130/80 mm Hg vs. 140-150/90 mm Hg will be applied from the time of randomization until delivery. Postpartum, clinicians will choose their own blood pressure goals as per JNC-7 guidelines.

Assessment of Outcomes:

For the pilot trial, maternal blood pressure is the primary outcome. This will be measured at weeks 20, 26, 32, 36 using a standardized method: after 15 minutes of rest, blood pressure will be measured with the woman seated, arm supported at heart level, bladder of cuff encircling >80% of arm circumference and phase V Korotkoff used for diastolic reading. Blood pressure will be recorded three times, five minutes apart, and the mean of these values will allow assessment of BP control in the study.

Secondary outcomes:

1. The incidence of superimposed preeclampsia in chronically hypertensive women. Diagnosis of superimposed preeclampsia will be made by the following criteria:

   * Worsening hypertension after 20 weeks
   * AND proteinuria >.3g/day on 24 hour collection when there was previously none OR doubling of proteinuria, in those positive at baseline
   * AND/OR the HELLP syndrome (hemolysis on blood smear, liver transaminase levels > 2 x normal, low platelets <100/mm3).
2. Gestational age
3. Birth weight < 10th centile for gestational age
4. Serious perinatal complications including neonatal death, respiratory distress, intraventricular hemorrhage, hypotension, bradycardia, and maternal complications of eclampsia, stroke, or end organ failure, cesarean section. Preterm admission, severe hypertension and indication for delivery will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant patients will be evaluated for recruitment to 13 6/7 weeks gestation.
2. Age 18-50
3. Patients will be included for consideration to enter this trial if office blood pressure is >140/90 mm Hg: systolic >140 mm Hg, diastolic >90 mm Hg or both. The average of 3 readings taken a minimum of 5 minutes apart will be recorded as the baseline blood pressure.
4. Patients will also be included for consideration to enter this trial if they have known longstanding hypertension DBP >90 within 2 years of index pregnancy and/or are on antihypertensive medication, regardless of in-office blood pressure if seen in their first trimester.

Exclusion Criteria:

Significant target organ damage; at the patient's initial antepartum visit, routine serum creatinine and urine dipstick for protein are performed by the attending obstetrician. If the patient has been hypertensive by history for over 5 years, a screening electrocardiogram will be performed. These will be reviewed for results precluding participation in the trial.

1. Known renal disease creatinine > 1.2 mg/dl
2. Proteinuria >500 mg/day at baseline
3. Left ventricular hypertrophy by ECG criteria.
4. History of the following: chronic illness requiring immunosuppression, as well as secondary causes of hypertension: pheochromocytoma, hyperaldosteronism, coarctation of aorta, renal artery stenosis not revascularized.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2004-07; Primary Completion 2005-03 (Actual); Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
The achievement of target blood pressure obtained at every six weeks visits: weeks 20, 26, 32 and 38

SECONDARY OUTCOMES:
The incidence of superimposed preeclampsia
Gestational age
Birth weight < 10th centile for gestational age
Serious perinatal complications

CONTACTS AND LOCATIONS:
Overall Officials: Phyllis August, MD MPH, Principal Investigator — The New York PresbyterianHospital-Weill Medical College of Cornell University
Locations (1):
- The New York PresbyterianHospital-Weill Medical College of Cornell University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Study terminated